CLINICAL TRIAL: NCT01386073
Title: Efficacy of FreshKote and Systane for the Treatment of Dry Eye and Improvement of Osmolarity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: Melissa Earl, CRO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Focus2011-001
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FreshKote (Active Comparator)
  Interventions: Drug: FreshKote
- Systane (Placebo Comparator)
  Interventions: Drug: Systane

INTERVENTIONS:
Drug: FreshKote — Three times a day for three months
  Arms: FreshKote
Drug: Systane — three times a day for three months
  Arms: Systane

SUMMARY:
The purpose of this study is to compare the efficacy of FreshKote and Systane for the reduction of dry eye signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye patients with Level 2 disease or greater as defined by the Delpi Panel
* Tear osmolarity of at least 308 mosm
* At least 18 years of age, Male or Female
* Willing to provide written informed consent
* Likely to complete all study visits
* If currently using ocular lubricants, must complete a 10-14 day washout

Exclusion Criteria:

* Presence of any active ocular disease other than dry eye
* Use of topical ophthalmic medications
* Use of contact lenses during the trial
* Pregnant or nursing, or planning a pregnancy. Patients will be asked if they are pregnant or may be pregnant and excluded if they answer in the affirmative.
* Any known sensitivity to any ingredients of either study drop
* Oral anti-inflammatory medications, omega 3 supplements, or doxycycline
* Punctal plugs inserted within the last 6 months or less
* Uncontrolled systemic disease
* Subjects with known sensitivity or inappropriate responsiveness to any of the medications used.
* Acute or chronic disease or illness that would increase risk or confound study results (e.g., uncontrolled diabetes mellitus, immunocompromised, etc.)
* Corneal abnormalities (e.g., ecstatic diseases, degenerations, or corneal dystrophies of the stroma or endothelium)
* Concurrent participation or participation in the last 30 days in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
TBUT | Three months
  Test that measures how long it takes for the tears to break up
Best Corrected Visual Acuity | Three months
  Vision obtained with the best possible lens correction (glasses or contact lenses)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pepose, MD, Principal Investigator — Pepose Vision Institute; Mitch Jackson, MD, Principal Investigator — Jackson Eye, S.C
Locations (2):
- United States (2):
  - Jackson Eye, S.C, Lake Villa, Illinois
  - Pepose Vision Institute, Chesterfield, Missouri